CLINICAL TRIAL: NCT00132964
Title: Randomized Control Trial of Casting Versus Ankle Bracing in Children With Low-risk Ankle Fractures
Brief Title: Brace Versus Casting in Pediatric Low Risk Ankle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Kathy Boutis, Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000000188
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Ankle Fracture
Keywords: pediatric; ankle fractures; randomized controlled trial; management
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immobilizaton device (Active Comparator): Below Knee walking cast
  Interventions: Device: Below knee walking cast
- Immobilization device (Experimental): Removable ankle brace
  Interventions: Device: Removable ankle brace

INTERVENTIONS:
Device: Below knee walking cast — Not required
  Arms: Immobilizaton device
Device: Removable ankle brace — not required
  Arms: Immobilization device

SUMMARY:
Acute ankle fractures are common in children. Most of these are stable and have a low risk of problems in the future. Even though these fractures are benign, these injuries are often casted for a fixed time period, which is inconvenient, expensive, and does not appear to be a practice that has been proven to be scientifically correct.

Therefore, in this study, in healthy children with low-risk ankle fractures, we, the investigators at the Hospital for Sick Children, will examine if a removable ankle brace is at least as good as casting with respect to how well and how fast children return to their usual activities. In addition, we will compare the costs of each method for the patient and the health care system.

Successful management of low-risk fractures with an ankle brace will allow for several advantages over the use of the cast. These advantages include the possibility of returning to normal activities faster, fewer visits to specialty hospital clinics, and significant cost savings.

DETAILED DESCRIPTION:
Objective: To determine if a removable ankle brace is at least as effective as casting in children between 5 and 18 years old with low-risk ankle fractures.

Rationale: Ankle injuries are very common among children. The Canadian Health Injury Reporting and Prevention Program reports approximately 5500 ankle injuries per year in children presenting to the 16 participating emergency departments, 35% of which are fractures. The majority of ankle injuries in children, including ankle fractures, have an excellent prognosis with a very low risk for any complications. We have recently shown that a predefined structured 'low-risk' clinical exam reliably identifies these low risk injuries, while simultaneously excluding 100% of high-risk fractures. This clinical rule reduces the need for radiography in children with ankle injuries by 63%. However, all low-risk injuries are currently not managed uniformly. Low-risk ankle fractures are often treated with a cast while soft tissue injuries are treated in a brace. Due to this distinction in management, many physicians still feel compelled to do radiographs in children with low risk ankle injuries in order to identify the fractures. We will now expand our previous work to show that all low risk ankle fractures can be safely treated in the same way as soft tissue injuries of the ankle. The current treatment of low risk fractures is casting which is inconvenient, necessitates orthopedic referral, and may be associated with soft tissue complications. Furthermore, casting is not an evidence-based practice. Preliminary evidence in adults with stable ankle fractures suggests that an ankle brace may offer a safe alternative to casting, while allowing comparable resumption of usual activities and less reliance on sub-specialty care. Therefore, the primary purpose of this study is to compare the functional outcomes that result from ankle bracing with those from casting in children with low-risk ankle fractures.

Design: In this randomized, outcomes assessor blinded, single center trial, children diagnosed with low-risk ankle fractures will receive either an ankle brace or a below-knee walking cast.

Outcome Measures: The primary outcome measure will be an assessment of functional daily activities as measured by the modified performance Activities Scale for Kids (ASKp) at four weeks post injury. Secondary outcomes will include an assessment of pain scores, ankle range of motion and return to baseline function. A concurrent health economic evaluation will be conducted using both patient and health care sector costs.

Sample Size and Analysis: The null hypothesis for the primary analysis is that the brace is less effective than casting by at least five percentage points on the ASKp scale. Assuming a standard deviation of 10%, alpha = 0.05, beta = 0.2 and 10% dropout rate yields a sample size of 112 patients. Secondary analyses will include Fisher's Exact test to compare proportions of children with full range of motion of the injured ankle at four weeks and with full baseline activity level at four months, and the area under the curve of a pain-time profile curve will be compared using a Student's t-test. An economic analysis will assess the incremental net benefit of bracing versus casting from a health care perspective.

Significance: If the removable brace is found to be at least as effective as the cast, this study has the potential to standardize the treatment of all low risk ankle injuries. Since these injuries can be reliably detected by physical examination, routine radiography of these injuries can be eliminated. These injuries could therefore be safely treated by primary physicians, thereby reducing the number of emergency department visits, obviating the need for orthopedic referral, or a return visit for cast removal. As a result, this study will provide critical information about the optimal treatment for the majority of ankle injuries in children from the perspective of clinical efficacy and health economics.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 18 years of age with one of the following fractures:

  * Undisplaced Salter-Harris types I and II fractures of the distal fibula;
  * Avulsion fractures of the distal fibula or distal fibular epiphysis;
  * Metaphyseal buckle fractures of the distal fibula;
  * Lateral talus fractures.

Exclusion Criteria:

* The diagnosis of ankle sprain or contusion; they occur primarily in adolescents with closed epiphyseal plates.
* All open fractures which require surgical debridement.
* All children at risk for pathological fractures such as those with congenital or acquired generalized bony disease.
* Congenital anomalies of the feet and/or ankles.
* Patients with coagulopathies.
* Multisystem trauma and multiple fractures of the same or opposite limb.
* Patients cognitively and developmentally delayed with inability to express pain and/or difficult assessment of baseline activity level.
* Injuries greater than 72 hours old.
* Past history of surgery or closed reduction of the same ankle within the last 6 months or ankle trauma of the same ankle within 3 months.
* Patients who do not have phone or electronic mail access.
* Patients living outside the Greater Toronto area (GTA) and who are unwilling to meet the physiotherapist at Hospital for Sick Children (HSC) for the four week assessment.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 2003-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy K Boutis, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Boutis K, Willan AR, Babyn P, Narayanan UG, Alman B, Schuh S. A randomized, controlled trial of a removable brace versus casting in children with low-risk ankle fractures. Pediatrics. 2007 Jun;119(6):e1256-63. doi: 10.1542/peds.2006-2958. PMID 17545357

RESULTS

PARTICIPANT FLOW:
Groups:
- Immobilizaton Device: Below Knee walking cast was placed on the ankle injury.
- Immobilization Device: Removable ankle brace was placed on the injured ankle.
Period: Overall Study
Arm/Group | Immobilizaton Device | Immobilization Device
Started | 54 | 57
Completed | 50 | 54
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immobilizaton Device | Immobilization Device | Total
Number analyzed (Participants) | 54 | 57 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54 | 57 | 111
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.55 (2.91) | 9.94 (2.43) | 10.2 (2.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 29 | 32 | 61
Region of Enrollment [Number; unit: participants]
  Canada | 54 | 57 | 111

OUTCOME MEASURES:

1. Primary Outcome: Functional Outcome as Measured by the Activities Scale for Kids at 4 Weeks From the Time of the Initial Injury
Description: Activities Scale for Kids (ASKp) measured by a physiotherapist at 4 week visit and is a validated 38-questionnaire that targets activities of children. The minimal scores are 0 and maximum are 100. Higher score indicates higher function.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: percentage of questions
Groups:
- Immobilization Device: Removable ankle brace that you placed on the injured ankle and can be removed as needed by the patient
Arm/Group | Immobilizaton Device | Immobilization Device
Number analyzed (Participants) | 50 | 54
percentage of questions | 85.3 (2.06) | 91.3 (1.14)

2. Secondary Outcome: Pain at 4 Weeks
Description: Bieri Face Pain Scale (BFPS). This is scored as 0, 2, 4, 6, 8, 10. The minimum and maximum values are 0 and 10 respectively. A higher score reports worse pain.
Time Frame: 4 weeks
Reporting Status: Not Posted, anticipated posting 2026-09

3. Secondary Outcome: Range of Motion at 4 Weeks
Description: Goniometer measured by a physiotherapist
Time Frame: 4 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Health Economic Outcomes
Description: parent reported costs and health care system costs
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Immobilizaton Device | Immobilization Device
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/57
Other Adverse Events (participants affected / at risk) | 4/54 | 16/57
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immobilizaton Device (N=54) | Immobilization Device (N=57)
Poor Fit of Immobilization Device (Skin and subcutaneous tissue disorders) | 4 (4) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes